CLINICAL TRIAL: NCT00544453
Title: Evaluation of [123I] MNI-308 and SPECT as a Marker of Beta-amyloid Protein Deposition in Subjects With Alzheimer Disease in Comparison to Healthy Subjects
Brief Title: Evaluation of [123I] MNI-308 and SPECT as a Marker of Beta-amyloid Protein Deposition in AD Subjects Compared to HC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Preliminary data showed [123I] MNI-308 not a useful tool in detection of AD.
Sponsor: Molecular NeuroImaging (Other)
Responsible Party: John Seibyl, MD; Senior Scientist, Institute for Neurodegenative Disorders
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MNI-308-01
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer Disease
Keywords: SPECT; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Iodine-123

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: [123I] MNI-308 — Injection of [123I] MNI-308 and SPECT scanning

SUMMARY:
The main objectives of this proposal are as follows:

To assess the dynamic uptake and washout of 123-I MNI-308, a potential imaging biomarker for β-amyloid burden in brain, using single photon emission computed tomography (SPECT) in similarly aged Alzheimer's (AD) subjects and healthy controls

To perform blood metabolite characterization of 123-I MNI-308 in healthy and AD subjects to determine the metabolic fate and nature of metabolites in assessment of 123-I MNI-308 as a single photon computed tomography (SPECT) brain imaging agent

Evaluate the test/retest reproducibility of 123-I MNI-308 and SPECT in AD subjects and healthy control

DETAILED DESCRIPTION:
General Design and Methods. The underlying goal of this study is to assess 123-I MNI-308 SPECT imaging as a tool to detect ß-amyloid deposition in the brain of AD research participants and age- and gender-matched healthy subjects. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. Approximately 10 patients with Alzheimers disease (AD) and 6 healthy controls (within +/- 2 years) will be recruited to participate in this study. Healthy controls will be examined to ensure that there is no evidence of neurodegenerative changes including cognitive decline.

An interval of at least 14 days will lapse between dosing in the first four AD subjects. This is intended to provide a longer period for AE assessments. Once complete, absent any serious adverse events in these initial AD subjects, dosing may commence with the remainder of the subjects, including healthy controls.

Informed consent will be obtained for all subjects. All subjects will undergo a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. Subjects will be asked to undergo a bolus injection of 123-I MNI-308. Subjects will undergo serial SPECT imaging scans and serial venous plasma sampling for measurement of 123-I MNI-308 in plasma (both protein bound and free) over a period of up to 8 hours. The imaging analyses will be performed by an image-processing specialist who will remain masked to the procedures employed with each imaging acquisition. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I MNI-308. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the AD patients and controls will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease will be recruited for this study. The following criteria will be met for inclusion of AD subjects in this study:

  * The participant is 50 years or older.
  * Written informed consent is obtained.
  * Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
  * Mini-Mental Status Exam score < 25.
  * Modified Hachinski Ischemia Scale score of ≤ 4.
  * Geriatric Depression Scales (GDS) ≤ 10.
  * For females, non-child bearing potential or negative urine or blood pregnancy test on day of 123-I MNI-308 injection.

Healthy Control Subject Selection. Healthy control subjects who have no neurological disease will be recruited for this study. The following criteria will be met for inclusion of healthy control subjects in this study:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* Mini-Mental Status Exam score ≥28.
* For females, non-child bearing potential or negative urine or blood pregnancy test on day of 123-I MNI-308 injection.

Exclusion Criteria:

* Alzheimer's subjects will be excluded from participation for the following reasons:

  * The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease.
  * The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
  * The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
  * The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Pregnancy

Healthy control subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danna L Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://www.indd.org